CLINICAL TRIAL: NCT03162913
Title: The Effects of Strawberry Supplementation on Memory and Gait Among Over-weight Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Human Nutrition Research Center on Aging (U.S. Federal Agency)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Principal Investigator, Barbara Shukitt-Hale, Research Psychologist, USDA Human Nutrition Research Center on Aging
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 12523
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Aging; Age-related Cognitive Decline; Obesity
Keywords: Strawberry; Cognition; Gait; Posture
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strawberry (Experimental): Participants randomized into this arm of the study consume freeze-dried strawberry powder.
  Interventions: Dietary Supplement: Strawberry
- Placebo (Placebo Comparator): Participants randomized into this arm of the study consume a strawberry placebo powder.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Strawberry — 12g freeze-dried strawberry (powder), twice daily with water, for 90 days
  Arms: Strawberry
Other: Placebo — 12g red, strawberry-flavored powder, twice daily with water, for 90 days
  Arms: Placebo

SUMMARY:
This study is being conducted to assess the effect of dietary strawberry supplementation on cognition and mobility in obese middle-aged and older adults. It is hypothesized that plant compounds, present in strawberries, may improve cognition and mobility.

DETAILED DESCRIPTION:
Previously, the investigators have shown that dietary berry fruit are able to reverse several parameters of brain aging, as well as age-related motor and cognitive deficits when fed to aged rats. They have shown that strawberry, in particular, can reduce oxidative stress and pro-inflammatory signaling in the brain and improve both mobility and cognition. A recent study also found that the addition of two servings of strawberry per day for 3 months could significantly improve verbal and spatial memory among healthy older adults, particularly on tests with high cognitive demand. These effects may reflect the direct effects of strawberries' bioactive and neuroavailable polyphenols on brain signaling or their indirect effects through antioxidant and anti-inflammatory pathways. However, participants in that study were selected from a healthy aging population, which made it difficult to detect changes in balance, mobility, and the less complex cognitive tasks. Therefore, the investigators are proposing the current study to assess the effects of dietary strawberry on mobility and cognition among a compromised population, obese older adults, who are at increased risk for cardiovascular, metabolic, and neurodegenerative disease. The risk for heart disease, diabetes, stroke, cancer and dementia increases in direct relation to overweight and obesity measures, and research now shows that obesity is a primary cause of mental deterioration among the middle-aged and senior populations. In this study, obese older adults (55-75yo, BMI 30-36) will consume 24g/d freeze-dried strawberry or control powder for 3 months and complete a battery of lifestyle, mobility, and cognitive tests at 3 time points. The investigators hypothesize that supplementing obese older adults' diet with strawberry will improve performance on complex tasks involving mobility and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 55 and 75 years
* Body mass index (BMI) between 30-40
* Hemoglobin A1C level between 5.7 and 6.4%
* Height between 60 and 74 inches tall
* Adequate visual acuity or corrected visual acuity to read and perform computer tasks
* Fluency in spoken and written English
* Ability to walk independently for 20 minutes as per self-report.
* Women must be postmenopausal (absence of menstruation for a minimum of 12-months or bilateral oophorectomy)
* Willing to abstain from recreational drug use

Exclusion Criteria:

* Vegetarian or vegan
* Cognitive impairment, memory loss, or neurologic/psychological disorder that interfere with activities of daily living
* Muscle or mobility deficit that would interfere with walking independent for 20 minutes
* Chronic conditions associated with increased risk of falls or falls within the last year that were not precipitated by unusual circumstances (e.g. slipping on ice, being pushed)
* Gastrointestinal diseases, conditions, or medications influencing gastrointestinal absorption
* Use of medications or dietary supplements known or suspected to influence study outcomes
* Mini Mental State Exam (MMSE) score of less than 24 at screening
* Diabetes mellitus diagnosis or fasting glucose >= 126 mg/dL or taking diabetes medication
* Liver dysfunction, history of cirrhosis, or elevated SGPT, SGOT, or total bilirubin
* Kidney disease as indicated by serum creatinine > 1.5 mg/dL at screening
* Uncontrolled blood pressure
* Cardiac or pulmonary conditions that limit ambulation or results in dyspnea with ambulation
* Allergy to strawberry or ingredients in the placebo.
* Ethanol use above 2 servings/day of beer (12-ounces), wine (5 ounces) or liquor (1.5 ounces), or binge-drinking
* Recent inflammatory diseases (for example: rheumatoid arthritis, lupus)
* Cigarette smoking, use of nicotine replacement products, or smoking of marijuana/consumption of edibles in past 3 months or during the course of the study
* History of stomach or bowel resection (other than appendectomy), gastric bypass or other bariatric weight loss procedure
* Cancer of any type (except for non-melanoma skin) in past 3 yrs or actively using cancer chemotherapeutic agents
* Clotting/bleeding disorders or ongoing anticoagulant use
* Bilateral mastectomy with nodal dissection
* No social security number (unable to pay stipend)
* Blood biochemistries outside of normal range
* Prior participation in a study involving berry supplementation at our institution

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Spatial Cognition | Change from baseline at 90 days
  Spatial cognition will be measured using a virtual navigation task.

SECONDARY OUTCOMES:
Gait Speed | Change from baseline at 90 days
  Preferred gait speed will be measured using an instrumented treadmill.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy M Scott, PhD, Principal Investigator — Tufts University; Barbara Shukitt-Hale, PhD, Principal Investigator — USDA Human Nutrition Research Center on Aging
Locations (1):
- Tammy M Scott, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller MG, Shukitt-Hale B. Berry fruit enhances beneficial signaling in the brain. J Agric Food Chem. 2012 Jun 13;60(23):5709-15. doi: 10.1021/jf2036033. Epub 2012 Feb 3. PMID 22264107
- [Background] Joseph JA, Shukitt-Hale B, Denisova NA, Bielinski D, Martin A, McEwen JJ, Bickford PC. Reversals of age-related declines in neuronal signal transduction, cognitive, and motor behavioral deficits with blueberry, spinach, or strawberry dietary supplementation. J Neurosci. 1999 Sep 15;19(18):8114-21. doi: 10.1523/JNEUROSCI.19-18-08114.1999. PMID 10479711
- [Background] Miller MG, Thangthaeng N, Poulose SM, Shukitt-Hale B. Role of fruits, nuts, and vegetables in maintaining cognitive health. Exp Gerontol. 2017 Aug;94:24-28. doi: 10.1016/j.exger.2016.12.014. Epub 2016 Dec 21. PMID 28011241
- [Background] Shukitt-Hale B, Bielinski DF, Lau FC, Willis LM, Carey AN, Joseph JA. The beneficial effects of berries on cognition, motor behaviour and neuronal function in ageing. Br J Nutr. 2015 Nov 28;114(10):1542-9. doi: 10.1017/S0007114515003451. Epub 2015 Sep 22. PMID 26392037
- See also: USDA Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University — http://hnrca.tufts.edu/
- See also: Agricultural Research Service (USDA) — http://www.ars.usda.gov/main/main.htm
- See also: California Strawberry Commission — http://www.calstrawberry.com/